CLINICAL TRIAL: NCT00873301
Title: The Effectiveness of Vestibulectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Prof. Jacob Bornstein, Chairman, Obstetrics and Gynecology, Western Galilee Hospital-Nahariya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JB 13-08-2008
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Vulvodynia
Keywords: vulvodynia; vestibulectomy; surgery; vestibulitis
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- vulvodynia (Experimental)
  Interventions: Procedure: vestibulectomy

INTERVENTIONS:
Procedure: vestibulectomy — Evaluation of the outcome of vestibulectomy which is the treatment of vulvar vestibulitis

SUMMARY:
Women with vulvodynia will fill out a questionnaire and undergo a gynecological examination before and 6 months after vestibulectomy. The investigators hypothesize that pain will decrease.

ELIGIBILITY:
Inclusion Criteria:

* vulvodynia, scheduled for vestibulectomy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
pain | 6 months following surgery

SECONDARY OUTCOMES:
sexual function | 6 months afater surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee Hospital- Nahariya, Nahariya, Israel